CLINICAL TRIAL: NCT07388472
Title: Retention and Caries-Preventive Outcomes of Glass Ionomer-Based Fissure Sealants in Children: A 24-Month Split-Mouth Randomized Controlled Trial
Brief Title: Glass Ionomer-Based Fissure Sealants in Children
Acronym: Sealant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ebru KUCUKYİLMAZ, Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014/100
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Fissure Sealant
Keywords: caries; prevention; glass ionomer material; fissure sealant

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double-blind, split-mouth design A total of 400 sealants were applied to the two fully erupted mandibular first molars of each participant. Following randomization, one molar received GC Fuji Triage (high-fluoride containing/control), while the contralateral molar received either GC Fuji VII EP (CPP-ACP-containing) or GCP Glass Seal (nano-fluorohydroxyapatite-containing).
Who Masked: Participant, Outcomes Assessor
Masking Description: The study was carried out as a double-blinded trial, whereby neither the patients nor the clinical evaluator was aware of what material was applied to each tooth. No blinding was done during the treatment period because all treatments were performed by one dentist. The randomization process was applied with two phases to ensure unbiased allocation of the fissure sealant materials to the participants. In the first phase of the randomization, which material groups (GC Fuji Triage -GCP Glass Seal/GC Fuji Triage-GC Fuji VII EP) would be applied to each patient was determined using a computer-generated randomization online tool (htpp//randomizer.org). In the second phase of the randomization, the allocation of the material to either the left or right mandibular molar of each participant was established through the coin toss method (heads or tails), and the opposing molar tooth was treated with the other material in accordance with the group designated by the first randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPP-ACP-containing fissure sealant (Experimental): In this group, one mandibular molar was treated with a high-fluoride glass ionomer-based fissure sealant (Fuji Triage, GC Corporation, Tokyo, Japan; control group), while the contralateral molar was treated with a CPP-ACP-containing fissure sealant (Fuji VII EP, GC Corporation, Tokyo, Japan)
  Interventions: Other: Retention of Fissure Sealants
- Nano-fluorohydroxyapatite-containing fissure sealant (Experimental): In this group, one mandibular molar was treated with a high-fluoride glass ionomer-based fissure sealant (Fuji Triage, GC Corporation, Tokyo, Japan; control group), while the contralateral molar was treated with nano-fluorohydroxyapatite-containing fissure sealant (GCP Glass Seal, GCP Dental, Vianen, The Netherlands)
  Interventions: Other: Retention of Fissure Sealants

INTERVENTIONS:
Other: Retention of Fissure Sealants — Other: Retention of the fissure sealants evaluated Description: Following classification system was employed for the retention evaluation of the sealants: 1 = complete retention; 2 = partial loss; or 3 = complete loss.

SUMMARY:
This study aimed to comparatively evaluate the 24-month clinical retention performance and caries-preventive efficacy of three glass ionomer-based fissure sealants with different compositions.

DETAILED DESCRIPTION:
This study aimed to comparatively evaluate the 24-month clinical retention performance and caries-preventive efficacy of three glass ionomer-based fissure sealants with different compositions.

This randomized, controlled, double-blind, split-mouth clinical trial was conducted with approval from the Medhical Ethics Committee of İzmir Kâtip Çelebi University (14/100) and registered at ClinicalTrials.gov (NCT07110701). The study included 200 healthy children (ASA I), aged 6-12 years, with moderate caries risk. A total of 400 sealants were applied to the two fully erupted mandibular first molars of each participant. Following randomization, one molar received GC Fuji Triage (high-fluoride containing/control), while the contralateral molar received either GC Fuji VII EP (CPP-ACP-containing) or GCP Glass Seal (nano-fluorohydroxyapatite-containing). Applications were performed by a single clinician in accordance with manufacturers' instructions. Patients were evaluated at 3-, 6-, 12-, 18-, and 24-months. Retention, marginal integrity, marginal discoloration, and secondary caries were assessed using modified USPHS criteria. Occlusal caries progression was monitored via ICDAS-II codes and DIAGNOdent measurements

ELIGIBILITY:
Inclusion Criteria:

* The study comprised 200 healthy children aged between 6 and 12 years, ASA class I (American Society of Anesthesiologists),
* 27 who were determined to exhibit cooperative behavior with a score of 3 or 4 on the Frankl Behavior Rating Scale.
* All participants had fully erupted lower first permanent molars on both sides which required the application of pit and fissure sealants.
* The inclusion criteria were based on the International Caries Detection and Assessment System II (ICDAS II) criteria,28 including deep and retained pits and fissures, no restorations, and no evidence of caries lesions.
* The teeth were examined using the caries diagnosis device (DIAGNOdent pen 2190, KaVo, USA); readings of ≤ 15 were included in the study as well.

Exclusion Criteria:

* Participants with special needs or systemic disease (ASA classification II or higher),
* requiring emergency dental care,
* suffering from a severe gag reflex or
* an allergy to latex,
* exhibiting uncooperative behavior (Frankl Score 1 or 2),
* exhibiting molars with anomalies of the enamel/dentin, or
* unable to attend follow-up appointments were excluded from the study.
* A bitewing radiograph was used to assess teeth suspected of having caries on their proximal surfaces, and those with caries were excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
retention rates of fissure sealants | The evaluation of pit-and-fissure sealants was conducted to record the presence of caries lesions and sealant retention at 6-, 12-, 18-, and 24 month follow-up visits.
  Following classification system was employed for the retention evaluation of the sealants: 1 = complete retention; 2 = partial loss; or 3 = complete loss.

CONTACTS AND LOCATIONS:
Overall Officials: EBRU KUCUKYİLMAZ, PROFESSOR, Study Chair — İZMİR KATIP CELEBI UNİVERSİTY
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study plan will be shared
Supporting Information: Study Protocol
Time Frame: The plan will be shared following the completion of the research paper (approximately 1 month)
Access Criteria: De-identified individual participant data (IPD) will be made available upon reasonable request following publication of the main results, in accordance with institutional and ethical regulations. Access will be granted to qualified researchers for non-commercial purposes.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT07388472/Prot_SAP_000.pdf